CLINICAL TRIAL: NCT06753240
Title: The Effects of Ultrasound-Guided Abdominal Plane Blocks on Postoperative Pain and Quality of Recovery in Laparoscopic Inguinal Hernia Repair
Brief Title: The Effects of Abdominal Plane Blocks on Postoperative Quality of Recovery
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İnan SARIDEDE, Research Assistant M.D in the Department of Anesthesiology and Reanimation, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH-INAN
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Laparoscopic Inguinal Hernia Repair; Quality of Recovery (QoR-15); Postoperative Analgesia; Regional Anesthesia
Keywords: laparoscopic inguinal hernia repair; m-tapa block; tap block; quality of recovery; patient controlled analgesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In laparoscopic inguinal hernia surgeries, although the effects of classical transversus abdominis plane (TAP) and Modified thoracoabdominal nerve block through perichondrial approach (m-TAPA) blocks on perioperative pain control and opioid consumption have been evaluated in various studies using classical scaling methods, their impact on postoperative recovery quality remains an area open for further research. In this observational study, the investigator's primary goal is to evaluate the effects of lateral approach TAP and m-TAPA blocks, which are routinely used for postoperative analgesia, on postoperative pain and recovery quality in patients undergoing laparoscopic inguinal hernia surgery, using the QoR-15 scale. The investigator's secondary goal is to contribute to identifying the standard analgesia method that will reduce postoperative opioid use, nausea, and vomiting, and improve recovery quality.

DETAILED DESCRIPTION:
Laparoscopic surgery is widely used in the repair of inguinal hernias, but it can cause moderate to severe postoperative pain. Perioperative pain management is essential for ensuring early mobilization of patients, reducing postoperative side effects and hospital stay durations, improving patient satisfaction, and preventing the development of chronic pain after surgery. The quality of postoperative recovery is influenced by various factors, such as the patient's preoperative characteristics, the type of surgery, the level of postoperative pain, and analgesic methods. In recent years, alongside traditional scales measuring classical parameters in evaluating postoperative recovery quality, new measurement tools focusing on patient satisfaction have been developed. One of these tools is the Quality of Recovery-15 (QoR-15) scale, which has been recommended by the European Society of Anaesthesiology for use in clinical studies investigating postoperative patient comfort and pain levels. This scale includes 15 questions across five different areas evaluating postoperative recovery from various perspectives: pain, physical comfort, physical independence, psychological support, and emotional state. The result is a score between 0 and 150, with higher scores indicating better recovery quality.

Ultrasound (USG)-guided abdominal plane blocks are an important part of multimodal analgesia due to their ease of application, ability to provide long-lasting postoperative analgesia, and potential to reduce opioid consumption. Various regional anesthesia techniques can be used for pain control following laparoscopic inguinal hernia repair surgeries (TransAbdominal Pre-Peritoneal approach-TAPP). Some of these techniques include the Transversus Abdominis Plane (TAP) block and the Perichondrial Approach Modified Thoracoabdominal Plane (m-TAPA) block. The TAP block is performed in the neurofascial plane between the internal oblique and transversus abdominis muscles, creating a dermatomal sensory block at the T6-L1 levels. It can be applied laterally, subcostally, or posteriorly. The Perichondrial Approach Modified Thoracoabdominal Plane (m-TAPA) block is used more recently in upper and lower abdominal surgeries to provide effective analgesia due to its wider dermatomal coverage. The m-TAPA block is performed under ultrasound guidance by injecting a local anesthetic between the costal cartilage and the transversus abdominis muscle, providing abdominal analgesia from T4-L1 along the anterior and lateral abdominal wall. Both TAP and m-TAPA blocks are regional analgesia techniques commonly applied in our daily practice after abdominal surgeries. The choice of regional anesthesia technique is determined based on the surgical region, type of surgery, and the experience of the anesthesia team.

This study includes 60 patients aged 18-65 years, classified in the American Society of Anesthesiologists (ASA) physical risk class I-III, who are scheduled to undergo elective laparoscopic inguinal hernia repair surgery under general anesthesia at the General Surgery Department of Fatih Sultan Mehmet Training and Research Hospital.Participants who are planning to receive M-TAPA block defines as Group M-TAPA, and those who receive lateral TAP block defines as Group TAP, with 30 patients in each group. After obtaining ethical approval on 14.12.2023, patients will be informed about the study procedure one day before surgery, and those who consent will sign an informed consent form. The QoR-15 questionnaire, used to assess anesthesia and surgical recovery quality, will be administered to patients preoperatively, 24 hours post-surgery, and on the 15th postoperative day. The results will be recorded for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo laparoscopic unilateral inguinal hernia surgery under general anesthesia in elective conditions, by the General Surgery clinic between January 10, 2024 and October 17, 2024
* Aged between 18-65 years, with a Body Mass Index (BMI) < 35 kg/m²,
* Having an American Society of Anesthesiologists (ASA) physical risk score of I-III,
* Patients who have given informed consent.

Exclusion Criteria:

* Patients who refuse to participate in the study
* Emergency surgeries
* Patients who will undergo recurrent or bilateral surgery
* Patients with a BMI ≥ 35 kg/m²
* Presence of local infection or hematoma at the application site
* Presence of coagulopathy
* History of known local anesthetic allergy or toxicity
* Patients with a history of hematological, renal, or hepatic diseases, or advanced respiratory or cardiac failure
* Patients with difficulty in cooperation, Alzheimer's, dementia, or psychiatric and neurological diseases
* Patients with a history of chronic analgesic use, chronic alcohol use, or substance addiction
* Patients who do not speak Turkish or have a language barrier

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo laparoscopic unilateral inguinal hernia surgery under general anesthesia in elective conditions.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Numeric Rate Score (NRS) | During the postoperative period, the NRS scores of patients in motion and at rest will be recorded at 0, 15, and 30 minutes, as well as at 2, 4, 6, 12, and 24 hours in the ward.
  NRS is a 0 to 10 scale that describes pain from good to worst.
Quality of recovery-15 (QoR-15) score | The QoR-15 questionnaire will be administered to participants before surgery, 24 hours after surgery, and on the 15th postoperative day.
  Quality of Recovery-15 (QoR-15) questionnaire, is used to measure anesthesia and surgical recovery quality

SECONDARY OUTCOMES:
Postoperative nausea and vomiting scale (PONV) | During the postoperative period, the nausea and vomiting scores of patients will be assessed at 0, 15, and 30 minutes, as well as at 2, 4, 6, 12, and 24 hours in the ward.
  PONV is a 0 to 4 scale that describes nausea and vomiting from good to worst.
Sedation score | During the postoperative period, the sedation scores of patients will be assessed at 0, 15, and 30 minutes, as well as at 2, 4, 6, 12, and 24 hours in the ward.
  Sedation score is a 0 to 3 scale that describes sedation from good to worst.
Pain Controlled Analgesia (PCA) | PACU 0,15, 30th minutes and postoperative 2, 4, 6, 12, 24th hours]
  PCA includes 200mg Tramadol/100 ml SF- no infusion, 5cc bolus, 15 minutes lock.

CONTACTS AND LOCATIONS:
Overall Officials: Oznur Demiroluk, Associate Professor, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Ciftci B, Gungor H, Alver S, Akin AN, Ozdenkaya Y, Tulgar S. Clinical Experience for Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) in Five Patients. Dermatomal Evaluation and Application of Different Volumes: A Case Series and Review of Literature. Turk J Anaesthesiol Reanim. 2023 Aug 18;51(4):354-357. doi: 10.4274/TJAR.2022.221042. PMID 37587679
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Selvi O, Azizoglu M, Temel G, Tulgar S, Chitneni A, Cinar EN, Ozer Z, Gurkan Y. Translation and Validation of the Turkish Version of the Quality of Postoperative Recovery Score QoR-15: A Multi-Centred Cohort Study. Turk J Anaesthesiol Reanim. 2022 Dec;50(6):443-448. doi: 10.5152/TJAR.2022.21417. PMID 36511494
- [Background] Alver S, Ciftci B, Gungor H, Golboyu BE, Ozdenkaya Y, Alici HA, Tulgar S. Efficacy of modified thoracoabdominal nerve block through perichondrial approach following laparoscopic inguinal hernia repair surgery: a randomized controlled trial. Braz J Anesthesiol. 2023 Sep-Oct;73(5):595-602. doi: 10.1016/j.bjane.2023.05.001. Epub 2023 May 16. PMID 37201747